CLINICAL TRIAL: NCT03358030
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of ISIS 416858 (IONIS-FXIRX, an Antisense Inhibitor of Factor XI), Administered Subcutaneously to Patients With End-Stage Renal Disease on Hemodialysis
Brief Title: A Study of ISIS 416858 Administered Subcutaneously to Participants With End-Stage Renal Disease (ESRD) on Hemodialysis
Acronym: EMERALD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ISIS 416858 CS5; 2017-002165-21 (EudraCT Number); NL62709.000.17 (Other: Central Committee on Research Involving Human Subjects (CCMO))
Record Dates: First submitted 2017-11-13; First posted 2017-11-30 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: End-stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — ISIS 416858; Riboflavin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo, subcutaneously, within 2 hours post-dialysis, once weekly from Week 1 (Day 1) through Week 26 of treatment period.
  Interventions: Drug: Placebo
- Cohort A: ISIS 416858, 200 mg (Experimental): Participants received ISIS 416858, 200 mg, subcutaneously, within 2 hours post-dialysis, once weekly from Week 1 (Day 1) through Week 26 of treatment period.
  Interventions: Drug: ISIS 416858
- Cohort B: ISIS 416858, 250 mg (Experimental): Participants received ISIS 416858, 250 mg, subcutaneously, within 2 hours post-dialysis, once weekly from Week 1 (Day 1) through Week 26 of treatment period.
  Interventions: Drug: ISIS 416858
- Cohort C: ISIS 416858, 300 mg (Experimental): Participants received ISIS 416858, 300 mg, subcutaneously, within 2 hours post-dialysis, once weekly from Week 1 (Day 1) through Week 26 of treatment period.
  Interventions: Drug: ISIS 416858

INTERVENTIONS:
Drug: ISIS 416858 — Subcutaneous injection
  Other Names: IONIS-FXIRx
  Arms: Cohort A: ISIS 416858, 200 mg; Cohort B: ISIS 416858, 250 mg; Cohort C: ISIS 416858, 300 mg
Drug: Placebo — Subcutaneous injection
  Other Names: 0.9% sterile saline; Riboflavin
  Arms: Placebo

SUMMARY:
Evaluation of safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of ISIS 416858 for up to 204 participants with ESRD receiving chronic hemodialysis as assessed by FXI activity reduction.

DETAILED DESCRIPTION:
Evaluation of safety, PK, and PD of ISIS 416858 (Dose # 1, Dose #2 and Dose #3 once weekly) as compared to placebo as assessed by FXI activity reduction.

ELIGIBILITY:
Inclusion Criteria:

• End stage renal disease maintained on outpatient hemodialysis at a healthcare center for > 3 months from screening with hemodialysis at least 3 times per week for a minimum of 9 hours per week of prescribed treatment time and plan to continue this throughout the study.

Exclusion Criteria:

* Participants with a history of major medical event (previous acute coronary syndrome, stroke or transient ischemic attack or systemic thromboembolic event) within 3 months of screening, major surgery within 3 months of screening, or new major physical examination finding except for documented atrial fibrillation
* Active bleeding within the past 3 months from screening or documented bleeding diathesis (excluding uremia), coagulopathy, or recent prolonged compression time at arteriovenous fistula
* Screening values of:

  * Platelet count < 150,000 cells per millimeter cube (cells/mm^3)
  * < 180,000 cells/mm^3 for platelet function/activation subgroup
  * International normalized ratio (INR) > 1.4
  * Activated partial thromboplastin time (aPTT) > upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x ULN
  * Total bilirubin > ULN
  * Factor XI (FXI) activity < 0.3 units per milliliter (U/mL)
* Malignancy within 5 years, except basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated. Participants with malignancies that have been treated with curative intent and which have no reoccurrence within 5 years may also be eligible if approved by Sponsor Medical Monitor.
* Within 6 months prior to screening, have any of the following:

  * More than 3 episodes of severe hypoglycemia requiring the assistance of another person to actively administer carbohydrate, glucagon or other resuscitative actions
  * One event of hypoglycemia in which the participant required hospitalization
  * Recurrent syncope and recurrent hypotension in the inter-dialytic period requiring intervention
* Planned major surgery in the next 6 months, including participants receiving kidney transplant or participants that anticipate changing dialysis modality (i.e. hemodialysis to peritoneal dialysis)
* Concomitant use of anticoagulant/antiplatelet agents (e.g., warfarin, dabigatran, rivaroxaban, clopidogrel) that may affect coagulation (except low dose aspirin (≤ 100 mg/day) during Treatment and Post-treatment Evaluation Periods is not allowed. Stable does of heparins during dialysis are permitted
* Uncontrolled hypertension as judged by the Investigator. Participants with a pre- or post-dialysis blood pressure (BP) that is > 180 millimeters of mercury (mmHg) on at least 3 of last 5 dialysis treatments.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Ionis Investigative Site, Santiago de Compostela, A Coruna
  - Ionis Investigative Site, Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 10 countries (Latvia, Netherlands, Spain, Austria, Belgium, Bulgaria, Czech Republic, Greece, Canada, and Russian Federation) from 26 December 2017 to 10 July 2019.
Pre-assignment Details: A total of 213 participants were enrolled and randomized in the study. Out of 213, 3 participants did not receive the study drug
Period: Overall Study
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg
Started | 53 | 53 | 55 | 52
Treated (Safety population: All participants randomized who have received at least 1 dose of the study drug.) | 53 | 53 | 54 | 50
Per-protocol (PP) Population | 49 | 45 | 43 | 35
Completed | 50 | 52 | 46 | 48
Not Completed | 3 | 1 | 9 | 4
Not completed — Adverse Event or Serious Adverse Event (SAE) | 2 | 0 | 5 | 1
Not completed — Ineligibility | 0 | 0 | 0 | 2
Not completed — Voluntary Withdrawal | 1 | 1 | 3 | 1
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg | Total
Number analyzed (Participants) | 53 | 53 | 54 | 50 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13) | 61 (14) | 63 (12) | 58 (14) | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 19 | 20 | 81
  Male | 34 | 30 | 35 | 30 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 6 | 5 | 12
  Not Hispanic or Latino | 52 | 53 | 48 | 45 | 198
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 0 | 3
  White | 52 | 51 | 50 | 49 | 202
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Bleeding (MB) and Clinically Relevant Non-Major Bleeding (CRNMB)
Description: MB was defined as one of the following: Fatal bleeding; symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular if in a major joint, or pericardial, or intramuscular with compartment syndrome, clinically overt bleeding leading to transfusion of greater than or equal to (>=) 2 units of packed red blood cells or whole blood or a fall in hemoglobin of 20 grams per liter (g/L) (1.24 millimoles per liter [mmol/L]) or more within 24 hours. CRNMB was defined as overt bleeding not meeting the criteria for MB but that resulted, in either medical examination, intervention, or had clinical consequences for a participant.
Time Frame: Up to Day 260
Population: Safety population included all randomized participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg
Number analyzed (Participants) | 53 | 53 | 54 | 50
Participants | 3 | 2 | 3 | 3

2. Other Pre Specified Outcome: Percent Change From Baseline in Activated Partial Thromboplastin Time (aPTT)
Time Frame: Baseline (Day 1) up to Day 260
Population: PP population: All participants, randomized without missing > 2 doses during the first 12 weeks or > 5 doses over the 26-week Treatment Period (TP) and did not have any major protocol violations that would have affected the interpretation/integrity of study results. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg
Number analyzed (Participants) | 49 | 45 | 43 | 35
percentage change
  Percent Change From Baseline at Day 5: number analyzed (Participants) | 48 | 44 | 43 | 35
  Percent Change From Baseline at Day 5 | -2.8 (23.1) | 9.3 (41.5) | -2.8 (19.2) | 0.7 (18.2)
  Percent Change From Baseline at Day 12: number analyzed (Participants) | 47 | 43 | 42 | 34
  Percent Change From Baseline at Day 12 | 1.4 (33.5) | 9.4 (25.9) | 0.8 (21.9) | 3.6 (19.5)
  Percent Change From Baseline at Day 15: number analyzed (Participants) | 49 | 45 | 42 | 35
  Percent Change From Baseline at Day 15 | 3.8 (47.7) | 7.5 (29.0) | 12.5 (39.8) | 12.5 (38.4)
  Percent Change From Baseline at Day 22: number analyzed (Participants) | 48 | 44 | 43 | 35
  Percent Change From Baseline at Day 22 | -0.6 (25.6) | 11.4 (38.1) | 8.4 (30.4) | 16.6 (32.0)
  Percent Change From Baseline at Day 29: number analyzed (Participants) | 47 | 45 | 42 | 35
  Percent Change From Baseline at Day 29 | -1.9 (23.8) | 11.0 (28.4) | 11.4 (30.7) | 18.8 (46.6)
  Percent Change From Baseline at Day 36: number analyzed (Participants) | 47 | 45 | 42 | 35
  Percent Change From Baseline at Day 36 | -3.1 (17.8) | 7.1 (18.2) | 13.2 (35.5) | 16.9 (21.0)
  Percent Change From Baseline at Day 50: number analyzed (Participants) | 49 | 44 | 43 | 33
  Percent Change From Baseline at Day 50 | 6.8 (46.9) | 24.1 (53.4) | 27.5 (42.4) | 24.3 (34.3)
  Percent Change From Baseline at Day 64: number analyzed (Participants) | 48 | 44 | 42 | 35
  Percent Change From Baseline at Day 64 | 6.0 (36.1) | 20.3 (25.8) | 29.9 (75.6) | 40.5 (53.7)
  Percent Change From Baseline at Day 78: number analyzed (Participants) | 46 | 45 | 42 | 35
  Percent Change From Baseline at Day 78 | 6.6 (49.5) | 27.9 (49.2) | 27.9 (38.6) | 42.9 (47.8)
  Percent Change From Baseline at Day 92: number analyzed (Participants) | 47 | 45 | 42 | 34
  Percent Change From Baseline at Day 92 | 9.5 (58.8) | 19.1 (27.1) | 52.5 (83.1) | 42.1 (57.2)
  Percent Change From Baseline at Day 106: number analyzed (Participants) | 49 | 45 | 42 | 34
  Percent Change From Baseline at Day 106 | 10.9 (70.7) | 38.9 (71.7) | 28.5 (46.1) | 44.8 (60.7)
  Percent Change From Baseline at Day 120: number analyzed (Participants) | 45 | 44 | 42 | 35
  Percent Change From Baseline at Day 120 | 2.6 (26.6) | 28.5 (43.1) | 22.5 (33.1) | 41.4 (49.4)
  Percent Change From Baseline at Day 134: number analyzed (Participants) | 49 | 43 | 43 | 34
  Percent Change From Baseline at Day 134 | -6.2 (16.0) | 42.9 (86.6) | 29.5 (49.8) | 50.1 (98.1)
  Percent Change From Baseline at Day 148: number analyzed (Participants) | 47 | 45 | 43 | 34
  Percent Change From Baseline at Day 148 | 1.0 (25.8) | 26.1 (28.7) | 34.0 (53.5) | 38.7 (61.5)
  Percent Change From Baseline at Day 162: number analyzed (Participants) | 49 | 44 | 41 | 33
  Percent Change From Baseline at Day 162 | -1.6 (17.1) | 27.6 (30.1) | 31.6 (39.3) | 33.3 (34.9)
  Percent Change From Baseline at Day 176: number analyzed (Participants) | 47 | 45 | 42 | 33
  Percent Change From Baseline at Day 176 | 3.7 (31.6) | 28.8 (35.0) | 36.3 (79.0) | 32.3 (34.6)
  Percent Change From Baseline at Day 190: number analyzed (Participants) | 44 | 44 | 42 | 33
  Percent Change From Baseline at Day 190 | -3.6 (12.5) | 38.3 (92.9) | 20.5 (31.6) | 23.5 (20.2)
  Percent Change From Baseline at Day 204: number analyzed (Participants) | 46 | 44 | 41 | 33
  Percent Change From Baseline at Day 204 | -0.4 (27.9) | 17.4 (39.3) | 13.3 (27.1) | 16.9 (32.1)
  Percent Change From Baseline at Day 218: number analyzed (Participants) | 47 | 44 | 41 | 34
  Percent Change From Baseline at Day 218 | -0.7 (26.4) | 13.1 (25.8) | 7.0 (24.6) | 13.2 (30.3)
  Percent Change From Baseline at Day 232: number analyzed (Participants) | 47 | 43 | 41 | 33
  Percent Change From Baseline at Day 232 | -0.7 (41.8) | 8.6 (24.0) | 16.8 (44.0) | 3.1 (14.8)
  Percent Change From Baseline at Day 246: number analyzed (Participants) | 46 | 42 | 38 | 34
  Percent Change From Baseline at Day 246 | -0.0 (44.2) | 10.0 (26.9) | 3.5 (25.2) | 3.6 (20.6)
  Percent Change From Baseline at Day 260: number analyzed (Participants) | 46 | 41 | 40 | 34
  Percent Change From Baseline at Day 260 | 2.3 (50.7) | 16.1 (54.4) | -2.9 (21.6) | 3.6 (30.1)
Statistical Analysis 1: Comparison: Cohort A: ISIS 416858, 200 mg; Day 12 through Day 260; Test type: Other; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Cohort B: ISIS 416858, 250 mg vs Cohort C: ISIS 416858, 300 mg; Day 15 through Day 232; Test type: Other; p < 0.05, ANOVA

3. Other Pre Specified Outcome: Percent Change From Baseline in Factor XI (FXI) Activity
Time Frame: Baseline (Day 1) up to Day 260
Population: PP population: All participants, randomized without missing > 2 doses during the first 12 weeks or > 5 doses over the 26-week TP and did not have any major protocol violations that would have affected the interpretation/integrity of study results. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg
Number analyzed (Participants) | 49 | 45 | 43 | 35
percentage change
  Percent Change From Baseline at Day 5: number analyzed (Participants) | 46 | 43 | 40 | 35
  Percent Change From Baseline at Day 5 | -0.6 (14.4) | 2.5 (24.6) | -0.0 (14.8) | -2.5 (18.3)
  Percent Change From Baseline at Day 12 | -1.9 (13.7) | -3.0 (17.3) | -8.8 (18.7) | -14.1 (16.1)
  Percent Change From Baseline at Day 15 | -0.6 (15.1) | -7.1 (16.2) | -14.0 (21.3) | -18.8 (17.3)
  Percent Change From Baseline at Day 22 | -3.7 (18.2) | -17.2 (16.2) | -22.7 (19.5) | -27.6 (19.3)
  Percent Change From Baseline at Day 29 | -3.3 (18.3) | -21.4 (16.9) | -31.5 (23.4) | -37.9 (18.5)
  Percent Change From Baseline at Day 36 | -6.0 (18.1) | -26.3 (18.4) | -37.3 (22.0) | -42.8 (17.9)
  Percent Change From Baseline at Day 50 | -3.2 (19.7) | -37.9 (22.2) | -48.1 (24.1) | -55.7 (20.6)
  Percent Change From Baseline at Day 64 | -4.5 (20.2) | -41.8 (20.1) | -55.1 (24.0) | -61.7 (20.3)
  Percent Change From Baseline at Day 78 | -8.1 (19.6) | -44.6 (20.9) | -56.4 (23.9) | -64.2 (19.5)
  Percent Change From Baseline at Day 92 | -6.2 (16.0) | -45.0 (21.6) | -60.2 (21.8) | -66.0 (19.0)
  Percent Change From Baseline at Day 106 | -6.6 (19.2) | -49.4 (20.4) | -58.1 (22.2) | -67.8 (18.4)
  Percent Change From Baseline at Day 120 | -0.8 (23.0) | -47.8 (20.3) | -57.2 (28.1) | -66.9 (17.6)
  Percent Change From Baseline at Day 134 | -1.3 (18.1) | -50.0 (19.1) | -57.0 (28.0) | -67.7 (19.7)
  Percent Change From Baseline at Day 148 | -4.3 (23.6) | -50.4 (17.5) | -59.2 (24.0) | -65.5 (20.0)
  Percent Change From Baseline at Day 162 | -3.1 (22.8) | -48.9 (21.5) | -60.0 (23.4) | -64.1 (24.5)
  Percent Change From Baseline at Day 176 | -4.1 (23.6) | -49.9 (24.8) | -61.1 (21.2) | -64.3 (17.4)
  Percent Change From Baseline at Day 190 | -2.7 (17.8) | -45.4 (28.9) | -55.2 (22.2) | -60.9 (19.6)
  Percent Change From Baseline at Day 204 | -1.8 (25.0) | -36.9 (28.7) | -48.2 (24.3) | -52.2 (22.1)
  Percent Change From Baseline at Day 218 | -5.6 (17.8) | -29.3 (20.7) | -37.4 (22.8) | -41.8 (24.2)
  Percent Change From Baseline at Day 232 | -0.7 (18.6) | -19.5 (24.7) | -28.0 (21.2) | -29.6 (25.2)
  Percent Change From Baseline at Day 246 | -2.6 (21.0) | -13.6 (27.6) | -20.7 (18.4) | -22.3 (24.0)
  Percent Change From Baseline at Day 260 | -3.8 (21.3) | -11.1 (25.0) | -15.3 (19.5) | -16.0 (22.1)
Statistical Analysis 1: Comparison: Cohort A: ISIS 416858, 200 mg; Day 15 through Day 176; Test type: Other; p < 0.05, Wilcoxon Rank Sum Test; Wilcoxon Rank Sum Test based on t approximation
Statistical Analysis 2: Comparison: Cohort B: ISIS 416858, 250 mg vs Cohort C: ISIS 416858, 300 mg; Day 12 through Day 176; Test type: Other; p < 0.05, Wilcoxon Rank Sum Test; Wilcoxon Rank Sum Test based on t approximation

4. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities Related to Platelet Count
Description: Participants were assessed based on pre-defined criteria in the protocol for platelet count abnormality: 100 - less than (<)140, 75 - <100, 50 - <75, 25 - <50 and < 25 thousands per cubic millimeter (K/mm^3) based on investigator's discretion.
Time Frame: Up to Day 260
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg
Number analyzed (Participants) | 53 | 53 | 54 | 50
Participants
  100 - <140 K/mm^3 | 9 | 21 | 20 | 21
  75 - <100 K/mm^3 | 2 | 2 | 6 | 7
  50 - <75 K/mm^3 | 0 | 0 | 4 | 0
  25 - <50 K/mm^3 | 0 | 0 | 1 | 1
  < 25 K/mm^3 | 0 | 0 | 1 | 1

5. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities - Alanine Transaminase (ALT) and Aspartate Aminotransferase (AST)
Description: Participants were assessed based on pre-defined criteria in protocol for abnormality in ALT and AST values: Confirmed ALT (serum glutamic pyruvic transaminase [SGPT]); greater than (>) 3*Upper limit of normal range (ULN), >5*ULN and confirmed AST (serum glutamic-oxaloacetic transaminase [SGOT]); >3*ULN and >5*ULN. A confirmed value was based on a consecutive lab value within 7 days of the initial value. If that value was in the same or worse category the initial value was confirmed. If the consecutive value was in a better category then the initial value was confirmed using the consecutive value category. If there were multiple results on the same day, no matter from the same lab vendor or different lab vendors, then the worst value was used in the analysis. Abnormality in laboratory parameter was based on investigator's discretion.
Time Frame: Up to Day 260
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg
Number analyzed (Participants) | 53 | 53 | 54 | 50
Participants
  ALT: >3*ULN, Confirmed | 0 | 0 | 1 | 0
  ALT: >5*ULN, Confirmed | 0 | 0 | 1 | 0
  AST: >3*ULN, Confirmed | 0 | 0 | 1 | 0
  AST: >5*ULN, Confirmed | 0 | 0 | 1 | 0

6. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Time Frame: Up to Day 260
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg
Number analyzed (Participants) | 53 | 53 | 54 | 50
Participants | 33 | 37 | 46 | 44

7. Other Pre Specified Outcome: Percent Change From Baseline in Factor XI (FXI) Antigen Levels
Time Frame: Baseline (Day 1) up to Day 260
Population: PP population: All participants, randomized without missing > 2 doses during first 12 weeks or > 5 doses over 26-week TP and did not have any major protocol violations that would have affected interpretation/integrity of study results. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg
Number analyzed (Participants) | 49 | 45 | 43 | 35
percentage change | 11.3 (27.0) | -3.4 (17.5) | -10.1 (21.8) | -13.9 (22.7)

ADVERSE EVENTS:
Time Frame: Up to Day 260
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Cohort A: ISIS 416858, 200 mg | Cohort B: ISIS 416858, 250 mg | Cohort C: ISIS 416858, 300 mg
All-Cause Mortality (participants affected / at risk) | 3/53 | 0/53 | 5/54 | 1/50
Serious Adverse Events (participants affected / at risk) | 10/53 | 6/53 | 20/54 | 13/50
Other Adverse Events (participants affected / at risk) | 25/53 | 27/53 | 35/54 | 39/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Cohort A: ISIS 416858, 200 mg (N=53) | Cohort B: ISIS 416858, 250 mg (N=54) | Cohort C: ISIS 416858, 300 mg (N=50)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Death (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arteriovenous fistula maturation failure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 3
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Idiopathic intracranial hypertension (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dry gangrene (Vascular disorders) | 0 | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Cohort A: ISIS 416858, 200 mg (N=53) | Cohort B: ISIS 416858, 250 mg (N=54) | Cohort C: ISIS 416858, 300 mg (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4 | 2 | 0
Injection site bruising (General disorders) | 1 | 2 | 3 | 4
Injection site discolouration (General disorders) | 0 | 1 | 2 | 3
Injection site erythema (General disorders) | 1 | 6 | 6 | 14
Injection site haematoma (General disorders) | 2 | 12 | 8 | 9
Injection site pain (General disorders) | 2 | 4 | 7 | 6
Injection site pruritus (General disorders) | 2 | 5 | 6 | 11
Pyrexia (General disorders) | 1 | 0 | 1 | 3
Bronchitis (Infections and infestations) | 4 | 2 | 1 | 3
Respiratory tract infection (Infections and infestations) | 6 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 3
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 3 | 3 | 4 | 6
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 5
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 2
Haemoglobin decreased (Investigations) | 0 | 3 | 2 | 1
Platelet count decreased (Investigations) | 0 | 0 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1
Headache (Nervous system disorders) | 4 | 3 | 2 | 5
Insomnia (Psychiatric disorders) | 3 | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 5
Hypertension (Vascular disorders) | 3 | 2 | 1 | 1
Hypotension (Vascular disorders) | 1 | 4 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT03358030/Prot_SAP_000.pdf